CLINICAL TRIAL: NCT04918069
Title: Single-blinded, Randomized Study of Capsaicin to Prevent Delayed Chemotherapy-induced Nausea and Vomiting
Brief Title: Capsaicin to Prevent Delayed Chemotherapy Induced Nausea and Vomiting (CapCIN)
Acronym: CapCIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Heber Rew Bright, Lecturer, Christian Medical College, Vellore, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11995
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Chemotherapy; Capsaicin; Nausea and Vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin (Experimental): 2g of 0.075% topical capsaicin ointment applied four times daily (preferably to the abdomen) for the first five days of chemotherapy
  Interventions: Drug: Capsaicin
- Placebo (Placebo Comparator): 2g of topical placebo ointment applied four times daily (preferably to the abdomen) for the first five days of chemotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin — Topical capsaicin ointment
  Arms: Capsaicin
Drug: Placebo — Topical placebo ointment
  Arms: Placebo

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) is one of the few most severe adverse effects of chemotherapy, which often panic patients undergoing cancer treatment. Though acute episodes of CINV are well controlled with pharmacologic agents, delayed CINV continues to present a treatment challenge.

Significant progress has been made over the past many years in discovering the pathophysiology of CINV. Primarily, three areas in the brain including central pattern generator (CPG), nucleus tractus solitarius (NTS) and area postrema (AP) are implicated in generating emetic reflex in all types of CINV (anticipatory, acute and delayed). The latter two areas NTS and AP are located at the caudal end of the fourth ventricle of brain which lies outside of the blood brain barrier and hence are stimulated by agents present in either blood and/or cerebrospinal fluid (CSF). Furthermore, NTS and AP are rich in muscarinic, dopamine, serotonin, neurokinin (NK1) and histamine receptors which are particularly important in delayed CINV. Clinical trials of antimuscarinic, antidopaminergic, antihistaminic drugs to prevent CINV have yielded inconclusive results except for olanzapine which is known to act on multiple receptors in NTS/AP. Only NK1 antagonists (e.g. aprepitant) which prevent substance P (SP) from binding to NK1 receptors have shown promising results and are clinically used to prevent delayed CINV. SP is a tachykinin peptide encoded by TAC1 (tachykinin precursor 1) gene and is found abundant in both peripheral and CNS. NK1 receptors in NTS/AP upon binding with SP will generate emetic reflex which will trigger delayed CINV. Though the topical analgesic drug capsaicin is reported to interfere with endogenous SP, its antiemetic potential in CINV has not been studied. This study intend to explore the antiemetic potential of capsaicin which is known to interfere with SP release in the GIT and CNS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult chemotherapy naïve patients of at least 18 years old
2. Diagnosed with a malignant disease and scheduled for highly emetogenic chemotherapy (as defined by NCCN guidelines v1.2019)
3. No concurrent radiotherapy or use of other antiemetic drugs except (dexamethasone, ondansetron/granisetron, and olanzapine)
4. Normal renal and hepatic function

Exclusion Criteria:

1. Pregnant or breast feeding
2. Contraindication for capsaicin or other medications in the study
3. Has ongoing nausea and/or vomiting of other etiology
4. History of anticipatory nausea and/or vomiting or has vomited/nauseated within 24 hours prior to the start of scheduled chemotherapy
5. Chronic alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Nausea | Within 15 days of chemotherapy
  Number of participants with chemotherapy-induced nausea that occurs after 24 hours of the first cycle
Vomiting | Within 15 days of chemotherapy
  Number of participants with chemotherapy-induced vomiting that occurs after 24 hours of the first cycle

SECONDARY OUTCOMES:
Overall chemotherapy-induced nausea and vomiting | Within 15 days of chemotherapy
  Number of participants with both immediate and delayed chemotherapy-induced nausea and vomiting
Severity of chemotherapy-induced nausea and vomiting | Within 15 days of chemotherapy
  Number of participants with severe, moderate and mild chemotherapy-induced nausea and vomiting
Use of rescue medication | Within 15 days of chemotherapy
  Number of participants requiring rescue medication for nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Heber Rew Bright, MPharm, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared depending on prevailing local institutional policies.

REFERENCES:
- [Derived] Bright HR, Singh A, Joel A, Georgy JT, John AO, Rajkumar P, Jiji H, Stehno-Bittel L, Samuel P, Chandy SJ. Randomized Placebo-Controlled Trial of Topical Capsaicin for Delayed Chemotherapy-Induced Nausea and Vomiting. JCO Glob Oncol. 2024 Jun;10:e2400130. doi: 10.1200/GO.24.00130. PMID 38905580